CLINICAL TRIAL: NCT06032104
Title: Feasibility of Pulses Supplementation in Healthy Adults: A Feeding Study
Brief Title: Feasibility and Colorectal Benefits of Pulses Supplementation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2012455
Record Dates: First submitted 2023-08-24; First posted 2023-09-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Polyp; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The randomized clinical trial has a cross-over design. The 20 participants will be randomized to a 14-day bean intervention versus usual care pre- or post-colonoscopy with a cross-over design. The 14-day bean intervention will be preceded by a 3-day ramp-up, acclimation, phase of beans feeding starting at one 1/2 cup of beans for day 1, followed by two 1/2 cups/day for days 2 and 3, then the full dose of three 1/2 cups/day for 14 days afterwards. Participants will be randomized 1:1 using a stratified randomization design. The randomization strata will be sex and presence/absence of metabolic syndrome factors with 1:1 ratio. Investigators anticipate a 20% dropout; therefore, investigators will recruit 25 participants to complete procedures on 20.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bean smoothie then usual diet (Experimental): Participants first receive 2 weeks of adding bean smoothie to usual diet before colonoscopy. After colonoscopy, they receive usual diet for 2 weeks
  Interventions: Dietary Supplement: Dry beans; Dietary Supplement: Usual diet
- Usual diet then bean smoothie (Experimental): Participants first receive 2 weeks of usual diet before colonoscopy. After colonoscopy, they add bean smoothie to usual diet for 2 weeks
  Interventions: Dietary Supplement: Dry beans; Dietary Supplement: Usual diet

INTERVENTIONS:
Dietary Supplement: Dry beans — 0.5 cup of Bush's Best Cannellini Beans, three times per day before meals blended into a smoothie. If interested and depending on tolerance, participants will also have the opportunity to gradually increase the bean smoothie to a maximum of 1 cup three times per day before meals during the last week of the two-week bean smoothie intervention. If patient cannot not tolerate 1.5 cup of canned cannellini bean, we will reduce per tolerance or offer the option of choosing a bean-based flour (100 gram/day, 23% fiber from Archer Daniels Midland)
Dietary Supplement: Usual diet — Usual diet without adding the bean smoothie

SUMMARY:
Beans are a forgotten staple food that shows promise in improving health. The goal of this study is to look at how bean supplementation affects metabolic and bowel health. In the long-term, the investigators believe this research will lead to a better understanding of the impact of beans on bowel health. The investigators also hope that this research study will help us understand ways to improve human diet and prevent colon cancer in the future.

DETAILED DESCRIPTION:
Investigators are seeking adults planning for a standard of care colonoscopies (part of the participant's usual care). As part of this feeding study, a participant will be randomly assigned to either two weeks of a dry bean smoothie that the investigators will provide in addition to the participant's usual diet or continue with participant's usual diet without the bean smoothie (including the food and drink guidelines for the colonoscopy) 2 weeks before or after the participant colonoscopy.

Participants' involvement in this research will also include 2 research visits plus a visit on the day of their scheduled standard-of-care colonoscopy (each research visit will be 30-60 minutes in length, scheduled close to 2-4 weeks prior to the colonoscopy, day of the colonoscopy, as well as 2-12 weeks after the colonoscopy, depending on participant availability. The investigators expect about 25 people aged 35-75 to participate in this research.

Participation in this study will involve collecting breath tests, fecal (stool) samples, 8 Teaspoons of blood, clinical data, and participant questionnaire data. At the time of colonoscopy, the investigators will also sample the mucosa lining of the bowel and remnant (leftover or discarded) tissue from an intestine biopsy obtained as part of the participant's clinical care. Participants will be asked to sign a separate HIPAA authorization form to allow the investigators to collect information from participant's medical records. This information will become part of the research data.

ELIGIBILITY:
Inclusions:

1. 30-80 years-old
2. Overweight or obesity (body mass index ≥ 25 kg/m2)
3. Planned for a standard of care colonoscopy for colon cancer screening

Exclusions:

1. Intolerance to a bean or high bean consumer based on a screening survey
2. Pregnancy or actively planning to get pregnant
3. Any active gastrointestinal disease resulting in disturbed gut function or malabsorption (e.g., chronic diarrhea or inflammatory bowel disease)
4. Current or history of any malignancy in the past 10 years.
5. Chronic use of opioids, anti-inflammatory drugs, antibiotics, prebiotics, or probiotics within 1 month of study endpoints
6. History of a significant systemic condition (e.g., heart disease, chronic kidney disease, liver dysfunction or immune suppression), or abnormal laboratory markers (e.g., abnormal liver enzymes, creatinine, clotting factors, or low platelets count). The severity of the intolerance to fiber/ the medical conditions/lab markers and eligibility will be defined after the careful interview of the patient/review of the medical records by Dr. Hussan)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Compliance with the bean smoothie intervention | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  Mean percentage completion of bean smoothie intervention and mean percentage with positive breath test over 2 weeks
Tolerance to the bean smoothie intervention | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  Compare the mean change in individual gastrointestinal symptoms and scores between paired baseline- and post- bean smoothie intervention vs. usual care. Patient-Reported Outcomes Measurement Information System (PROMIS) survey T sore range is 1-100, normal average T score is 50 (Standard deviation of 10).
Effect of the bean smoothie intervention on serum biomarkers of health | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  Compare the percent with abnormal complete metabolic panel or complete blood count between paired baseline- and post- bean smoothie intervention vs. usual care
Change in fecal abundance of microbiome genes with bean smoothie intervention | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  Fecal microbiome assessment using 16s/metagenomics assay. Investigators will compare the change in paired baseline- and post- bean smoothie intervention vs. usual diet
Change from baseline in the fecal and serum metabolome with bean smoothie intervention | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  Fecal and serum metabolomic assessment using an untargeted metabolomics assay. Investigators will compare the change in paired baseline- and post- bean smoothie intervention vs. usual diet
Impact of bean intervention on colonic tissue RNA markers of health | 2-4 weeks prior to colonoscopy till colonoscopy
  Compare colonic tissue RNA-seq assay between participants randomized to bean intervention vs usual care before the colonoscopy

SECONDARY OUTCOMES:
Change from baseline in body composition | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  Body fat and muscle percentage measured using bio impedance analysis (BIA). Investigators will compare the change in paired baseline- and post- bean smoothie intervention vs. usual diet
Change from baseline in body mass index (BMI) | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  BMI measured using standard techniques. Investigators will compare the change in paired baseline- and post- bean smoothie intervention vs. usual diet
Change from baseline in waist circumference | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  Waist circumference measured using standard techniques. Investigators will compare the change in paired baseline- and post- bean smoothie intervention vs. usual diet
Reported change from baseline in fitness level | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  Investigators will compare the mean change in Abadie Perceived Physical Fitness Scale between paired baseline- and post- bean smoothie intervention vs. usual care. Perceived Physical Fitness Scale score range is 12-60, normal mean score is 42.46
Reported change from baseline in and exercise per week | 2-4 weeks prior to colonoscopy, till 2-12 weeks after colonoscopy
  Investigators will use the modified Leisure-Time Exercise Questionnaire to compare the mean change in average weekly exercise (minutes of exercise per week) between paired baseline- and post- bean smoothie intervention vs. usual care

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Hussan, MD, Principal Investigator — UC Davis
Locations (1):
- University of California Davis, Sacramento, California, United States